CLINICAL TRIAL: NCT04151043
Title: Analgesic Effects of Expectation and Deep Brain Stimulation in Patients With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: UAarhus_Sophie
Record Dates: First submitted 2019-10-28; First posted 2019-11-05 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-03

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Suggestion; Deep Brain Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Verbal suggestion (Other)
  Interventions: Behavioral: Suggestions; Device: Deep brain stimulation
- No suggestion (Other)
  Interventions: Behavioral: Suggestions; Device: Deep brain stimulation

INTERVENTIONS:
Behavioral: Suggestions — Verbal suggestions or no suggestions about treatment outcome
Device: Deep brain stimulation — Regulation of deep brain stimulation intensity

SUMMARY:
The study investigates analgesic effects of expectations and deep brain stimulation on chronic and evoked pain in patients with Parkinson's disease.

The study includes patients with Parkinson's disease that are exposed to pain stimuli through injection of hypertonic saline. During pain induction and chronic pain evaluation deep brain stimulation treatment is regulated. Pain stimuli and regulation of deep brain stimulation are accompanied by verbal suggestions as to the analgesic effect of deep brain stimulation or no suggestions. During the test session patients evaluate their chronic and evoked pain and expectations.

The study procedure is repeated on two separate test days to investigate pain during deep brain stimulation treatment with or without verbal suggestions. All participants will complete all study conditions with no suggestions and verbal suggestions, respectively.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of PD (confirmed by a neurologist)
* Bilateral implanted DBS in the STN during the study or for a minimum of 6 months

Exclusion criteria

* Other neurological or medical disorders (e.g. stroke, neuropathy, diabetes) or other disorders (e.g. musculoskeletal diseases) with expected influence on pain
* Dementia
* Untreated depression
* Patients unable to pause anti-parkinsonian medication
* Patients unable to cooperate
* Patients treated with painkillers except paracetamol and NSAID (except if pain and treatment is adequately stable as evaluated by a doctor)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Numerical rating scale (NRS) (Change) | Participants will be tested on two days. The numerical rating scale will be applied to assess chronic and evoked pain at baseline and in the five study conditions (after each deep brain stimulation regulation) on each day.
  A numerical rating scale from 0 (no pain) to 10 (worst pain) will be used to assess participants' subjective chronic and evoked pain in all study conditions.
Numerical rating scale (NRS) (Change) | Participants will be tested on two days. The numerical rating scale will be applied to assess expectations to chronic and evoked pain at baseline and in the five study conditions (after each deep brain stimulation regulation) on each day.
  A numerical rating scale from 0 (no pain) to 10 (worst pain) will be used to assess participants' subjective expectations to chronic and evoked pain in all study conditions.

SECONDARY OUTCOMES:
Unified Parkinson's Disease Rating Scale (UPDRS) (Change) | Participants will be tested on two days. The Unified Parkinson's Disease Rating Scale will be used to evaluate motor symptoms at baseline and in the five study conditions (after each deep brain stimulation regulation) on each day.
  Motor symptoms related to Parkinson's disease are assessed using the Unified Parkinson's Disease Rating Scale, part III in all study conditions.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychology and Behavioural Sciences, Aarhus University, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No